CLINICAL TRIAL: NCT04375618
Title: Efficacy of Recombinant Human Epidermal Growth Factor (RhEGF) Incorporated in An Absorbable Collagen Membrane for The Management of Gingival Recession Defects
Brief Title: RhEGF Incorporated in An Absorbable Collagen Membrane for The Management Of Gingival Recession Defects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVSIDS/perio/5/2019
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Periodontitis
Keywords: epidermal growth factor; gingival recession
MeSH Terms: conditions — Periodontitis; Gingival Recession | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGF impregnated in collagen membrane (Experimental): EGF impregnated in collagen membrane is placed in gingival recession defects
  Interventions: Drug: RhEGF
- plain collagen membrane (Active Comparator): plain collagen membrane is placed in gingival recession defects
  Interventions: Drug: Plain Collagen

INTERVENTIONS:
Drug: RhEGF — The EGF impregnated membrane will be placed upon the recession site and will be stabilized by suturing it to the lingual papillae using 4-0 absorbable sutures. The flap will be coronally advanced as far as possible to cover the membrane and will be sutured to the buccal interdental papillae with 4-0 absorbable sutures (Trulenetm, Healthium Medtech Pvt Ltd, Bangalore, India). Standard recall and maintenance regimen will be followed and subjects will be encouraged to report to the department on a monthly basis.
  Other Names: EGF+Collagen
  Arms: EGF impregnated in collagen membrane
Drug: Plain Collagen — A collagen membrane without FGF-2 will be used.
  Other Names: Control group
  Arms: plain collagen membrane

SUMMARY:
A sulcular incision will be made through each recession area and the tissues will be gradually undermined including the base of the interdental papilla. At the recession sites rhEGF incorporated absorbable collagen membrane will be gradually manipulated into the pouch through the tunnel till it covers the recession sites and will be stabilized with sutures.

DETAILED DESCRIPTION:
IN TEST SITE :

Local anesthesia will be administered and Vertical incisions will be given at interdental papillae away from recession defect site and a pouch will be created. A sulcular incision will be made through each recession area and the tissues will be gradually undermined including the base of the interdental papilla. At the recession sites rhEGF incorporated absorbable collagen membrane will be gradually manipulated into the pouch through the tunnel till it covers the recession sites and will be stabilized with sutures.

IN CONTROL SITE:

Same procedure will be done as the test site but plain collagen membrane will be gradually manipulated into the pouch through the tunnel till it covers the recession sites and will be stabilized with sutures.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male and female patients of age 20-55 yrs with Millers class I or class II gingival recession are included in the study.

Exclusion Criteria:

* Patients who are medically compromised and Subjects who underwent radiotherapy or chemotherapy and who are Smokers are excluded from the study

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Recession depth (RD) | Base line to 6months.
  Recession depth (RD) - measured from cementoenamel junction to most apical extension of gingival margin.

SECONDARY OUTCOMES:
Width of keratinized gingiva (KGW) | Base line to 6months.
  Width of keratinized gingiva (KGW) - distance between gingival margin and mucogingival junction will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- R V Chandra, Hyderabad, Telangana, India